CLINICAL TRIAL: NCT05346627
Title: Video Consultation and Mitochondrial Myopathies: Study of Efficacy and Tolerance of a Personalized Training Program at Home
Brief Title: Home Based Personalized Training and Video Consultation in Mitochondrial Myopathies: Study of Efficacy and Tolerance.
Acronym: TELE-MIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-GIRCI-01
Record Dates: First submitted 2022-04-08; First posted 2022-04-26 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Mitochondrial Myopathies
MeSH Terms: conditions — Mitochondrial Myopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mitochondrial myopathy (Other): Patient affected by mitochondrial myopathy, with genetic confirmation of mitochondrial DNA mutation
  Interventions: Procedure: Personalized and mixed training program

INTERVENTIONS:
Procedure: Personalized and mixed training program — Patients perform a personalized and mixed training program (endurance and muscle reinforcement), at home

SUMMARY:
Positive effect of physical activity on health arouses a strong interest at international level and is developped within the scope of national programs. Recommandations exist but must be designed for patients with functional limitations of activities.

Patients with mitochondrial diseases have exercice intolerance with an increase of muscular weakness and fatigue after low exercice volume. Theses patients have functional limitations of activities. In order to establish an appropriate training programme, it will be important to define and consider the physical condition. The Society of Mitochondrial Medecine published recommandations for management of theses patients,However, theses recommandations do not allow them to propose a training program of what can be done. For these vulnerable patients, therapists are responsible fo advising a training programm without guidelines to establish its terms and conditions. In addition, some exercices do not appear to have been the subject of complete assessmeents.

Regarding training programs (aerobic training, muscle reinforcement, miwed training), scientific literature shows a significant genetic and clinical variabilities, as well as a lack of data on clinical severity of included patients. In addition, the lack of informations regarding training effects of heteroplamy level limits our comprehension of mechanisms involved in adaptation of mitochondrial pool during training. Therefore, further reserchs on this subject are essential.

It is necessary to offer these patients a follow-up and personalized training program, which are in adequation with daily life. Some publications call on specifics concepts which are not compatible with day-to-day life. The investigators think it will be useful to investigate training effects in order to have practival conclusions, easily reproducible at home by patients with simple and inexpensive equipment. In this context, video consultation could allow the close follow-up of these patients.

The investigators hypothesize that a mixed training (endurance and muscle reinforcement), personalized, at home and followed by video consultation have positive effects on some physical criteria (such as musclar strength, tolerance to effort, functional abilities) without increasing heteroplasmy and creatine phosphokinase levels.

ELIGIBILITY:
Inclusion criteria:

* patient over 18 years-old,
* with genetically-confirmed mitochondria myopathy,
* with mitochondrial DNA mutation,
* clinically dominant myopathic-like disorders according investigator,
* able to walk with or without assistance,
* likely to be followed for at least one year without interruption by video consultation (implying internet connexion with computer and camera or smartophone),
* having given the written and informed consent and being social security member.
* For patients in childbearing age, she must have used at least one month if reliable contraception.

Exclusion criteria:

* patient wih pathology or comorbidity incompatible with the conduct of the study according the investigator during inclusion visit,
* patient with physical condition incompatible with training program according investigator during inclusion visit,
* patient having a physical tiredness and/or myalgia during last week with an intensity of 6 on visual and analog scale,
* pregnant or nursing patient,
* patient expecting pregnancy during the course of the study,
* patient protected by law or under guardianship or curatorship, or not able to participate in a clinical trial under L.1121-16 article of French Public Health Regulations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change of overall functional capacity of moving during training period from 6 months (S0) to 9 (S12) and 12 (S24) months | At 6 (S0), 9 (S12) and 12 (S24) months
  The overall functional capacity of moving will be measured by the time to perform the Timed Up and Go test.

SECONDARY OUTCOMES:
Change of muscular strength of upper and lower limbs during training period from 6 months (S0) to 9 (S12) and 12 (S24) months | At 6 (S0), 9 (S12) and 12 (S24) months
  Muscular strength of upper (shoulder abduction, elbow and fingers bending) and lower (knee extension) limbs during isometric and maximal muscular contractions will be measured with a quantified muscle testing device. Upper limbs strength will also measured during the developped sitting with dumbbells.
Change of muscular endurance of upper and lower limbs during training period from 6 months (S0) to 9 (S12) and 12 (S24) months | At 6 (S0), 9 (S12) and 12 (S24) months
  Muscular endurance of upper (shoulder abduction, elbow and fingers bending) and lower (knee extension) limbs during isometric and maximal muscular contractions, keeped during 30 secondes will be measured by the difference of the force between the beggining and the end of the contraction
Change of functional abilities in walking during training period from 6 months (S0) to 9 (S12) and 12 (S24) months | At 6 (S0), 9 (S12) and 12 (S24) months
  Modification of functional abilities in walking will be measured by the maximal distance of walking (in meter) during a 6-minutes walking test
Change of functional abilities during transferts during training period from 6 months (S0) to 9 (S12) and 12 (S24) months | At 6 (S0), 9 (S12) and 12 (S24) months
  Modification of functional abilities during transferts will be measured by the maximal number of transferts sitting to standing performed during a 1-minute chair lifts test
Change of clinical severity of the disease during training period from 6 months (S0) to 9 (S12) and 12 (S24) months | At 6 (S0), 9 (S12) and 12 (S24) months
  Clinical severity of the disease will be measured with the Newcastle Mitochondrial Disease Scale for Adults (NMDAS) and its 3 first sections. Score ranges from 0 to 145. The higher the score the more severe the disease.
Change of quality of life during training period from 6 months (S0) to 9 (S12) and 12 (S24) months | At 6 (S0), 9 (S12) and 12 (S24) months
  Quality of life will be measured with the Quality of Life in Genetic Neuromuscular Disease Questionnaire (QOL-gNMD). The QoL-gNMD is splitted in 3 domains: "Impact of Physical Symptoms" (score from 0 to 19), "Self-perception" (score from 0 to 24) and "Activities and Social Participation" (score from 0 to 27).
Change of tiredness felt during training period from 6 months (S0) to 9 (S12) and 12 (S24) months | At 6 (S0), 9 (S12) and 12 (S24) months
  The tiredness felt will be measured with the Fatigue Severity Scale (FSS). The FSS is a unidimensional scale which focuses on the physical aspects of fatigue. It is a self-reported questionnaire developed to measure the impact of disabling fatigue on daily functioning. It covers several areas including physical, social, and cognitive effects. The FSS is a patient-reported outcome composed of 9-items with scores ranging from 1 = "strongly disagree" to 7 = "strongly agree".
Check effects of a training program on clinical and biological tolerance, by assessing the modification of heteroplasmy level | At 6 (S0), 9 (S12) and 12 (S24) months
  Heteroplasmy level of mitochondrial DNA from blood and urine samples will be compared between the beginning of the training (6 months, S0), and 9 (S12) and 6 (S24) months after training period.
Check effects of a training program on clinical and biological tolerance, by regularly assessing the effort-related myalgia | From 6 months (S0) to 12 months (S24)
  Muscular pain level will be measured with the visual and analog scale for pain before and after each training session. Scorer ranges from 0 to 10, 0 being "no pain" and 10 being "maximum thinkable pain"
Check effects of a training program on clinical and biological tolerance, by assessing the blood creatine phosphokinase levels which is a muscle damage marker | From 0 (S-24) to 12 months (S24)
  Clinical and biological tolerance will be measured with the blood creatine phosphokinase levels before training and during training period (12 weeks before the begining of training period, at the begining of training period and 2, 4, 8, 12, 16, 20 and 24 weeks after the begining of training period)
Establish a "dose-effect" relationship between the training frequency and effects on clinical parameters (strength, endurance and functionnal abilities such as global moving, walking and during transferts) | From 0 (S-24) to 12 months (S24)
  Evolution of clinical markers (strength, endurance, global functional abilities in walking and during transferts) will be matched with number of completed training sessions, in order to identify a dose-effect relationship
Check effect of a training program on reported physical condition by assessing the Recent Physical Activity Questionnaire (RPAQ). | At 6 (S0), 9 (S12) and 12 (S24) months
  RPAQ is a splited in 3 parts: physical activity within and around the house, travel to and from work and your work activity and hobbies. This questionnaire assess:
  * physical activity level (inactive if score is less than 8.3 Metabolic Equivalent of Task (MET).h/week, moderate if score ranges from 8.3 to 16.7 MET.h/week or high physical activity if score is greater than 16.7 MET.h/week)
  * sedentary time (settled is score is greater than 7 hours per day or not settled if score is less than or equal to 7 hours per day).
Check effect of a training program on reported physical condition by assessing the Global Physical Activity Questionnaire (GPAQ). | At 6 (S0), 9 (S12) and 12 (S24) months
  GPAQ is a splited in 3 parts: activities at work, to move from one place to another and hobbies. For each part, score is ranked according to 3 levels: low, moderate and intense.
Describe the natural history of disease without training on heteroplasmy level | At 0 (S-24) and 6 months (S0)
  Heteroplasmy level of mitochondrial DNA from blood and urine samples will be assessed at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0).
Describe the natural history of disease without training on blood creatine phosphokinase levels | At 0 (S-24) and 6 months (S0)
  Blood creatine phosphokinase levels will be assessed at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0).
Describe the natural history of disease without training on muscular strength of upper and lower limbs | At 0 (S-24) and 6 months (S0)
  Muscular strength of upper (shoulder abduction, elbow and fingers bending) and lower (knee extension) limbs during isometric and maximal muscular contractions will be measured with a quantified muscle testing device at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0). Upper limbs strength will also measured during the developped sitting with dumbbells at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0).
Describe the natural history of disease without training on functional abilities in walking | At 0 (S-24) and 6 months (S0)
  Modification of functional abilities in walking will be measured by the maximal distance of walking (in meter) during a 6-minutes walking test, at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0).
Describe the natural history of disease without training on functional abilities during transfert | At 0 (S-24) and 6 months (S0)
  Modification of functional abilities during transferts will be measured by the maximal number of transferts sitting to standing performed during a 1-minute chair lifts test, at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0).
Describe the natural history of disease without training on quality of life | At 0 (S-24) and 6 months (S0)
  Quality of life will be measured with the Quality of Life in Genetic Neuromuscular Disease Questionnaire (QOL-gNMD) at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0). The QoL-gNMD is splitted in 3 domains: "Impact of Physical Symptoms" (score from 0 to 19), "Self-perception" (score from 0 to 24) and "Activities and Social Participation" (score from 0 to 27).
Describe the natural history of disease without training on tiredness felt | At 0 (S-24) and 6 months (S0)
  The tiredness felt will be measured with the Fatigue Severity Scale (FSS), at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0). The FSS is a unidimensional scale which focuses on the physical aspects of fatigue. It is a self-reported questionnaire developed to measure the impact of disabling fatigue on daily functioning. It covers several areas including physical, social, and cognitive effects. The FSS is a patient-reported outcome composed of 9-items with scores ranging from 1 = "strongly disagree" to 7 = "strongly agree".
Describe the natural history of disease without training on reported physical condition by assessing the Recent Physical Activity Questionnaire (RPAQ). | At 0 (S-24) and 6 months (S0)
  RPAQ is a splited in 3 parts: physical activity within and around the house, travel to and from work and your work activity and hobbies. This questionnaire assess, at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0):
  * physical activity level (inactive if score is less than 8.3 Metabolic Equivalent of Task (MET).h/week, moderate if score ranges from 8.3 to 16.7 MET.h/week or high physical activity if score is greater than 16.7 MET.h/week)
  * sedentary time (settled is score is greater than 7 hours per day or not settled if score is less than or equal to 7 hours per day).
Describe the natural history of disease without training on reported physical condition by assessing the Global Physical Activity Questionnaire (GPAQ). | At 0 (S-24) and 6 months (S0)
  GPAQ is a splited in 3 parts: activities at work, to move from one place to another and hobbies. For each part, score is ranked according to 3 levels: low, moderate and intense. GPAC will be assessed at the beginning of observation phase (S-24) and 6 months later, at the beginning of the training (S0).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, Alpes Maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided